CLINICAL TRIAL: NCT01355068
Title: An Open Label, Randomized, Single Dose, Crossover Pivotal Bioequivalence Study of Epanutin Infatabs 50 mg (Sourced From Germany) Verses Dilantin Infatabs 50 mg (Sourced From Australia) in Healthy Subjects
Brief Title: A Study to Assess if Epanutin Infatabs 50 mg From Germany Are Similar to Dilantin Infatabs 50 mg From Australia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A4121010
Record Dates: First submitted 2011-05-12; First posted 2011-05-17 (Estimated); Results first posted 2011-12-14 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2011-11

CONDITIONS: Healthy
Keywords: phenytoin; chewable tablets; dilantin; epanutin; infatabs; bioequivalence; Partial seizure; Tonic-clonic seizure
MeSH Terms: conditions — Seizures | interventions — Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Active Comparator): Epanutin Infatabs 50 mg (sourced from Germany), 1 x 50 mg (REFERENCE)
  Interventions: Drug: Epanutin Infatabs (Phenytoin)
- Treatment B (Experimental): Dilantin Infatabs 50 mg (sourced from Australia), 1 x 50 mg (TEST)
  Interventions: Drug: Dilantin Infatabs (Phenytoin)

INTERVENTIONS:
Drug: Epanutin Infatabs (Phenytoin) — Chewable Tablet, 50 mg, Single dose
  Arms: Treatment A
Drug: Dilantin Infatabs (Phenytoin) — Chewable Tablet, 50 mg, Single dose
  Arms: Treatment B

SUMMARY:
In this study, the bioequivalence of Epanutin Infatabs® 50 mg (sourced from Germany) and Dilantin Infatabs® 50 mg (sourced from Australia) will be assessed. This is intended to be a pivotal bioequivalence study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years, inclusive.
* An informed consent document signed and dated by the subject.

Exclusion Criteria:

* Evidence or history of clinically significant abnormalities.
* Any condition possibly affecting drug absorption (e.g. gastrectomy).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4121010&StudyName=A%20Study%20to%20Assess%20if%20Epanutin%20Infatabs%2050%20mg%20from%20Germany%20Are%20Similar%20to%20Dilantin%20Infatabs%2050%20mg%20from%20Australia

RESULTS

PARTICIPANT FLOW:
Groups:
- Epanutin Infatabs 50 mg First, Then Dilantin Infatabs 50 mg: Single oral dose of Epanutin (phenytoin) infatabs 50 milligram (mg) chewable tablet in first intervention period; and single oral dose of Dilantin (phenytoin) infatabs 50 mg chewable tablet in second intervention period. A washout period of at least 7 days was maintained between each period.
- Dilantin Infatabs 50 mg First, Then Epanutin Infatabs 50 mg: Single oral dose of Dilantin (phenytoin) infatabs 50 mg chewable tablet in first intervention period; and single oral dose of Epanutin (phenytoin) infatabs 50 mg chewable tablet in second intervention period. A washout period of at least 7 days was maintained between each period.
Period: First Intervention Period
Arm/Group | Epanutin Infatabs 50 mg First, Then Dilantin Infatabs 50 mg | Dilantin Infatabs 50 mg First, Then Epanutin Infatabs 50 mg
Started | 13 | 13
Completed | 13 | 11
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout Period (at Least 7 Days)
Arm/Group | Epanutin Infatabs 50 mg First, Then Dilantin Infatabs 50 mg | Dilantin Infatabs 50 mg First, Then Epanutin Infatabs 50 mg
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | Epanutin Infatabs 50 mg First, Then Dilantin Infatabs 50 mg | Dilantin Infatabs 50 mg First, Then Epanutin Infatabs 50 mg
Started | 13 | 11
Completed | 13 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes participants randomized to receive Epanutin (phenytoin) infatabs 50 mg first and Dilantin (phenytoin) infatabs 50 mg first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (AUClast).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, and 72 hours (hrs) post-dose
Population: Pharmacokinetic (PK) parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Epanutin Infatabs 50 mg: Single oral dose of Epanutin (phenytoin) infatabs 50 mg chewable tablet (Reference) in either first intervention period or second intervention period.
- Dilantin Infatabs 50 mg: Single oral dose of Dilantin (phenytoin) infatabs 50 mg chewable tablet (Test) in either first intervention period or second intervention period.
Arm/Group | Epanutin Infatabs 50 mg | Dilantin Infatabs 50 mg
Number analyzed (Participants) | 24 | 26
ng*hr/mL | 21380.0 (6043.0) | 21370.0 (5571.2)
Statistical Analysis 1: Comparison: Epanutin Infatabs 50 mg vs Dilantin Infatabs 50 mg; Natural log transformed AUClast was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 101.33, 90% CI 2-sided [97.85 to 104.94]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hrs post-dose
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Epanutin Infatabs 50 mg | Dilantin Infatabs 50 mg
Number analyzed (Participants) | 24 | 26
ng/mL | 952.10 (229.25) | 976.50 (214.78)
Statistical Analysis 1: Comparison: Epanutin Infatabs 50 mg vs Dilantin Infatabs 50 mg; Natural log transformed Cmax was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 102.20, 90% CI 2-sided [97.18 to 107.47]

3. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC [0-∞])
Description: AUC (0-∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-t) plus AUC (t-∞).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hrs post-dose
Population: PK parameter analysis population included all randomized and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period. Here, the 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Epanutin Infatabs 50 mg | Dilantin Infatabs 50 mg
Number analyzed (Participants) | 23 | 25
ng*hr/mL | 21730.0 (6345.9) | 21740.0 (5816.7)
Statistical Analysis 1: Comparison: Epanutin Infatabs 50 mg vs Dilantin Infatabs 50 mg; Natural log transformed AUC (0-∞) was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 101.43, 90% CI 2-sided [97.56 to 105.47]

4. Secondary Outcome: Extrapolated Area Under the Curve (AUC Percent [%] Extrap)
Description: AUC%extrap is the percentage of AUC [0-∞] obtained by forward extrapolation. It is calculated as (AUC [0-∞] minus AUClast)*100/ AUC [0-∞], where AUC [0-∞] = Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0-∞) and AUClast is area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hrs post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Percent AUC
Arm/Group | Epanutin Infatabs 50 mg | Dilantin Infatabs 50 mg
Number analyzed (Participants) | 24 | 26
Percent AUC | 3.321 (4.884) | 3.198 (4.805)

5. Secondary Outcome: Plasma Decay Half Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hrs post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Epanutin Infatabs 50 mg | Dilantin Infatabs 50 mg
Number analyzed (Participants) | 23 | 26
hr | 14.380 (3.247) | 14.970 (4.777)

6. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hrs post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Epanutin Infatabs 50 mg | Dilantin Infatabs 50 mg
Number analyzed (Participants) | 24 | 26
hr | 3.51 [1.00 to 5.00] | 4.00 [1.00 to 6.00]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Epanutin Infatabs 50 mg | Dilantin Infatabs 50 mg
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 4/24 | 2/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epanutin Infatabs 50 mg (N=24) | Dilantin Infatabs 50 mg (N=26)
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.